CLINICAL TRIAL: NCT00891566
Title: Prolonged Versus Conventional Immobilization After Arthroscopic Repair for Medium to Large Size Rotator Cuff Tear. A Prospective Randomized Controlled Trial
Brief Title: Duration of Immobilization After Rotator Cuff Repair: Its Clinical Impact
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jae Chul Yoo, Samsung Medical Center
Other Study IDs: 2008-04-051
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Rotator Cuff Tear
Keywords: medium to large tear; rotator cuff tear; arthroscopic repair; repair integrity; immobilization
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Immobilization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Immobilization — compared the healing status for 8 weeks of immobilization with the conventional 4 weeks of immobilization after rotator cuff repair

SUMMARY:
The purpose of this study is to determine whether the immobilization period is helpful for the better healing of repaired rotator cuff.

The investigators hypothesis is that the longer immobilization after rotator cuff repair will help the healing of rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* Medium to large sized cuff tear (2-4 cm)
* Yes subscapular partial fraying or longitudinal split side to side
* Yes acromioplasty
* Yes AC arthritis with mumford procedure
* Yes biceps tenotomy or tenodesis

Exclusion Criteria:

* No arthritic changes of glenohumeral joint
* No combined infection
* No mini-open procedures
* No complete subscapularis tear
* No incomplete repair
* No small tears or side to side repairs without anchors
* No pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: medium to large size rotator cuff tears
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
repair integrity analysis using postoperative MRI | 6 months

SECONDARY OUTCOMES:
American Shoulder and Elbow Surgeons' score | 2 year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Pennekamp W, Gekle C, Nicolas V, Seybold D. [Initial results of shoulder MRI in external rotation after primary shoulder dislocation and after immobilization in external rotation]. Rofo. 2006 Apr;178(4):410-5. doi: 10.1055/s-2006-926476. German. PMID 16607589
- [Result] Lewis CW, Schlegel TF, Hawkins RJ, James SP, Turner AS. The effect of immobilization on rotator cuff healing using modified Mason-Allen stitches: a biomechanical study in sheep. Biomed Sci Instrum. 2001;37:263-8. PMID 11347400
- [Result] Kim SH, Yoo JC, Ahn JM. Arthroscopically repaired Bankart lesions and the effect of two different arm positions on immediate postoperative evaluation with magnetic resonance arthrography. Arthroscopy. 2005 Jul;21(7):867-74. doi: 10.1016/j.arthro.2005.04.109. PMID 16012501
- [Derived] Koh KH, Lim TK, Shon MS, Park YE, Lee SW, Yoo JC. Effect of immobilization without passive exercise after rotator cuff repair: randomized clinical trial comparing four and eight weeks of immobilization. J Bone Joint Surg Am. 2014 Mar 19;96(6):e44. doi: 10.2106/JBJS.L.01741. PMID 24647511